CLINICAL TRIAL: NCT06619431
Title: Rumbo: an Integrated Mobile and Web-Based Application to Overcome Barriers to Receive Substance Use Disorder (SUD) Treatment and Improve Outcomes for Spanish-Speaking, Hispanic and Latinx Individuals
Brief Title: Pilot Test of a Mobile App That Helps Spanish-speakers Find Mental Health Services in the US.
Status: Completed | Type: Observational
Sponsor: Volver Health (Industry)
Collaborators: Boston University (Other); Pacific Institute for Research and Evaluation (Other); National Institute on Drug Abuse (NIDA) (NIH); National Institute on Drug Abuse (NIDA) (DA038095) (Unknown)
Responsible Party: Sponsor
Other Study IDs: R43DA057759 (NIH); 1R43DA057759-01 (NIH)
Record Dates: First submitted 2024-09-16; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Health Disparity, Minority and Vulnerable Populations
Keywords: Consumer health informatics; Health Disparities; Treatment access for hispanics/latinos

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Focus Group: The group consisted of three subgroups of Spanish-speakers: women, men, and caretakers.
  Interventions: Device: Mobile Application

INTERVENTIONS:
Device: Mobile Application — "Rumbo" is an easily shared bi-lingual application that helps Hispanic individuals with unhealthy substance use find and access treatment services and related resources. The application stands out from other eHealth tools by leveraging the collective efficacy of the Hispanic community to overcome barriers and support individuals' self-efficacy for engaging the treatment system. Rumbo's simple, user-centered design provides less-acculturated Hispanic individuals with a culturally appropriate tool to understand their needs within the complex US treatment system. Rumbo is comprised of four innovations: (1) a sharing function that facilitates its own implementation among the target population; (2) culturally responsive content and design; (3) problem identification and treatment navigation enhanced to include related resources; (4) an API that is designed for interoperability across extant technologies.

SUMMARY:
The goal of this observational study is to develop and test a mobile app for Spanish speakers residing in the US who seeking drug treatment and/or behavioral health services for themselves or an associate. The main questions it aims to answer are:

What are the features and content needed on this app?

How will people use and share this app?

Will they connect with treatment services?

After receiving input from focus group participants and other community stakeholders, the app was made available and its usage was tracked to determine its long-term, broad-scale feasibility.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Identify as Hispanic/Latino
* Own a smartphone, pad, or computer
* Be willing to meet with study personnel more than once

Exclusion Criteria:

* Age less than 18 or more than 75
* Evidence of significant cognitive impairment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hispanic/Latine community sample
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-04-02 (Actual); Study Completion 2024-04-02 (Actual)

PRIMARY OUTCOMES:
System Usability Scale | From enrollment to the close of end-user testing after 4 weeks.
  The system usability scale (SUS) is a ten-item attitude scale giving a global view of subjective assessments of usability.

CONTACTS AND LOCATIONS:
Overall Officials: William P Campbell, Principal Investigator — Volver Health
Locations (1):
- Volver Health, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: Yes
Data from participants will be reported when the study is published ion a peer-reviewed journal.
Supporting Information: Study Protocol
Time Frame: Upon publication in the Spring of 2025, and available indefinitely after that.
Access Criteria: Anyone with access to academic journals may access the data. Also, anyone may write to the study authors to receive a free copy of the published report.

REFERENCES:
- See also: Website of Volver Health, who conducted the study. — https://volver.health